CLINICAL TRIAL: NCT06931587
Title: Methyl Alcohol Intoxication as a Public Health Issue: A 3-Year Retrospective Analysis
Brief Title: Methanol Poisoning
Status: Completed | Type: Observational
Sponsor: Kartal City Hospital (Other)
Responsible Party: Principal Investigator, AKIN BİLİR, Medical Doctor, Kartal City Hospital
Other Study IDs: Kartal City Hospital
Record Dates: First submitted 2025-04-03; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Methanol Poisoning
Keywords: methanol; intoxication; Intensive care; mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study addresses methyl alcohol intoxications with profound acidosis requiring intensive care treatment. The goal is to contribute both to the improvement of diagnosis and follow-up processes and to the development of management strategies under the highlight of existing literature.

This study is a single-center, retrospective, observational cohort study conducted on patients admitted to the ICU between January 2022 and March 2025 with suspected or laboratory-confirmed methyl alcohol intoxication. The investigators analyzed patients' demographic characteristics, prognostic clinical and laboratory parameters, treatment approaches and outcomes

DETAILED DESCRIPTION:
This study addresses methyl alcohol intoxications with profound acidosis requiring intensive care treatment. The objective is to contribute to the improvement of diagnostic and follow-up processes, as well as to the development of management strategies, in light of the existing literature.

The study is a single-center, retrospective, observational cohort analysis conducted on patients admitted to the intensive care unit (ICU) between January 2022 and March 2025 with suspected or laboratory-confirmed methyl alcohol intoxication.

Data collection was performed in three steps. Initially, the hospital's electronic medical database was searched using the ICD code T51.1 to identify relevant cases. Subsequently, detailed medical records were reviewed to assess clinical progress and treatment interventions. Finally, laboratory findings were obtained through the hospital's patient record system.

Demographic characteristics-including age and gender-reasons for ICU admission, pre-existing conditions, presenting symptoms, and disease severity based on Acute Physiology and Chronic Health Evaluation II (APACHE II), Glasgow Coma Scale (GCS), Sequential Organ Failure Assessment (SOFA), and Simplified Acute Physiology Score (SAPS) evaluated during the first 24 hours of ICU stay were retrospectively analyzed. Treatment interventions, including ethanol or fomepizole administration, the need for hemodialysis (intermittent hemodialysis [IHD] or continuous venovenous hemodialysis [CVVHD]), supportive therapies, ICU length of stay, and clinical outcomes were also documented.

Laboratory evaluations included arterial blood gas analysis, anion gap, osmolality, complete blood count, glucose, urea, creatinine, electrolytes (sodium, potassium, chloride), C-reactive protein (CRP), and organ function tests such as aspartate aminotransferase (AST) and alanine aminotransferase (ALT).

Demographic data, prognostic clinical and laboratory parameters, treatment modalities, and clinical outcomes were analyzed by the investigators.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of methyl alcohol intoxication.

Exclusion Criteria:

* Other toxic alcohol intoxications
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes patients admitted to the ICU between January 2022 and March 2025 with suspected or laboratory-confirmed methyl alcohol intoxication.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
ICU Mortality Among Patients With Methyl Alcohol Intoxication | Up to 30 days (during ICU follow-up)
  Mortality was defined as death occurring during ICU stay among patients admitted with laboratory-confirmed or suspected methyl alcohol intoxication.

CONTACTS AND LOCATIONS:
Overall Officials: banu çevik, professor doctor, Study Chair — Kartal Dr. Lütfi Kirdar City Hospital
Locations (1):
- Kartal Dr. Lütfi Kırdar City Hospital, Kartal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all
Supporting Information: Study Protocol
Time Frame: 5/4/2025-5/4/2026

REFERENCES:
- [Background] Alhusain F, Alshalhoub M, Homaid MB, Esba LCA, Alghafees M, Al Deeb M. Clinical presentation and management of methanol poisoning outbreaks in Riyadh, Saudi Arabia: a retrospective analysis. BMC Emerg Med. 2024 Apr 16;24(1):64. doi: 10.1186/s12873-024-00976-1. PMID 38627622

DOCUMENTS (2):
  • Study Protocol (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT06931587/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT06931587/SAP_001.pdf